CLINICAL TRIAL: NCT00480805
Title: HYZAAR Versus Ramipril Diabetic Patients
Brief Title: HYZAAR vs. Ramipril for Diabetes (0954A-245)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-245; 2007_554
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Losartan; Hydrochlorothiazide; hydrochlorothiazide, losartan drug combination; Duration of Therapy

INTERVENTIONS:
Drug: MK0954A, losartan potassium (+) hydrochlorothiazide (HYZAAR) / Duration of Treatment : 8 Weeks
Drug: Comparator : ramipril /Duration of Treatment : 8 Weeks

SUMMARY:
A study to test the safety and efficacy of HYZAAR as compared to Ramipril in patients with type 2 diabetes mellitus (high blood sugar) and hypertension (high blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old, has been diagnosed with type 2 diabetes mellitus

Exclusion Criteria:

* Patient has renal disease, malignant hypertension, uncontrolled type 2 diabetes mellitus, history of stroke, TIA (Transient Ischemic Attacks) , or heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2001-08-08 (Actual); Primary Completion 2002-10-15 (Actual); Study Completion 2002-10-16 (Actual)

PRIMARY OUTCOMES:
To determine the antihypertensive effectiveness of HYZAAR as compared to Ramipril as measure by SiSBP at Week 4

SECONDARY OUTCOMES:
To determine the safety anf tolerability of HYZAAR as compared to Ramipril as seen in overall adverse experiences for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Fox JC, Leight K, Sutradhar SC, Demopoulos LA, Gleim GW, Lewin AJ, Bakris GL. The JNC 7 approach compared to conventional treatment in diabetic patients with hypertension: a double-blind trial of initial monotherapy vs. combination therapy. J Clin Hypertens (Greenwich). 2004 Aug;6(8):437-42; quiz 443-4. doi: 10.1111/j.1524-6175.2004.03488.x. PMID 15308882